CLINICAL TRIAL: NCT04932161
Title: Comparative Efficacy of Titanium Granules Over Hydroxyapatite in the Treatment of Periodontal Intrabony Defects: A Clinico-radiographic Study
Brief Title: Efficacy of Titanium Granules in the Treatment of Periodontal Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/4/2020
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Intrabony Periodontal Defect
Keywords: Intrabony defects; Titanium Granules
MeSH Terms: interventions — Durapatite

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium Granules as a bone graft in intrabony defects (Experimental): In test group, after reflection of flap and degranulation, bone graft i.e., titanium particles will be placed in the void created by the defect and sutures will be placed.
  Interventions: Procedure: Titanium Granules
- Hydroxyapatite as a bone graft in intrabony defects (Active Comparator): In control group, after reflection of flap and degranulation, bone graft i.e., hydroxyapatite will be placed in the defect and sutures will be placed.
  Interventions: Procedure: Hydroxyapatite

INTERVENTIONS:
Procedure: Titanium Granules — After degranulation of the intrabony defect, titanium particles will be placed in the defect and will be sutured.
  Arms: Titanium Granules as a bone graft in intrabony defects
Procedure: Hydroxyapatite — After degranulation of the intrabony defect, hydroxyapatite will be placed in the defect and will be sutured.
  Arms: Hydroxyapatite as a bone graft in intrabony defects

SUMMARY:
The ideal goal of the periodontal treatment is not only to prevent the progression of the disease, but also the regeneration and reconstruction of lost tissues. Many surgical techniques have been used to regenerate intrabony defects (IBD).

Titanium stimulates activation of the complement system, surface binding of platelets, and platelet activation as reflected by increased levels of platelet-derived growth factor, which is a substantial promoter of bone growth. Hence we may speculate that using a bone substitute made of titanium may be positive from the perspective of bone formation in osseous defects.

DETAILED DESCRIPTION:
Titanium granules consist of irregular porous granules of commercially pure titanium. The porous properties may lead to ingrowth of newly formed bone.The osseointegrating response to titanium may be the result of the potent activation of the intrinsic coagulation system and the subsequent release of growth factors from platelets.Therefore, the aim of this study is to compare the effect of titanium particles and hydroxyapatite on osseous regeneration in intrabony defects.

After reflection of flap and degranulation, bone graft i.e., titanium particles (test group) or hydroxyapatite(control group) will be placed in the void created by the defect and sutures will be placed.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy male and female patients of age >18 years with two-walled or three-walled intrabony defects and probing pocket depths (PPD) of >3mm.

Exclusion Criteria:

Medically compromised patients, patients <18 years of age, pregnant women, heavy smokers, and patients who underwent radiotherapy or chemotherapy are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | from baseline to 6 months
  Assessment of clinical attachment level using UNC-15 probe at baseline and post operatively at 3 and 6 months.
Probing Depth | from baseline to 6 months
  Assessment of probing depth using University of North Carolina(UNC)-15 probe at baseline and postoperatively at 3 and 6 months.
Bone Regeneration | at 3 months and 6 months
  Radiovisiography (RVG) will be used to assess bone regeneration achieved post operatively after 3 months and 6 months.

SECONDARY OUTCOMES:
Plaque Index | from baseline to 6 months
  Assessment of plaque (PI) - according to Turesky modification of Quigley and Hein Plaque Index, 1970.
Gingivitis | from baseline to 6 months
  Assessment of Gingivitis (GI) - according to Loe H and Silness P, 1963.

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Telangana, India